CLINICAL TRIAL: NCT00901511
Title: Inhaled GM-CSF Reduces the Need for Whole Lung Lavage and Improves Gas Exchange in Autoimmune PAP Patients
Brief Title: Inhaled GM-CSF Therapy of Autoimmune PAP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Collaborators: Agenzia Italiana del Farmaco (Other Government)
Responsible Party: Principal Investigator, Ilaria Campo, Study coordinator, Fondazione IRCCS Policlinico San Matteo di Pavia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FARM7MCPK4; Codice Interno 19900508; EudraCT 2008-007086-23
Record Dates: First submitted 2009-05-11; First posted 2009-05-13 (Estimated); Results first posted 2023-06-26 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Autoimmune Pulmonary Alveolar Proteinosis
Keywords: Whole lung lavage; GM-CSF; Sargramostim; aPAP
MeSH Terms: conditions — Pulmonary Alveolar Proteinosis, Acquired | interventions — sargramostim; Macrophage Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- GM-CSF Group (Experimental): Scheduled Baseline WLL: All participants will receive scheduled bilateral WLL at baseline (month 0).
  GM-CSF induction treatment: All participants will receive inhaled GM-CSF (250 mcg daily, 7 consecutive days every other week for 12 weeks beginning 1 week after the scheduled baseline WLL).
  Washout period: All participants will not receive inhaled GM-CSF treatment for 4 weeks immediately following GM-CSF induction treatment.
  GM-CSF maintenance treatment: All participants will receive inhaled GM-CSF (250 mcg daily on days 1 and 3 of every consecutive 14-day period for 6 months beginning 17 weeks after the scheduled baseline WLL).
  Unscheduled Rescue WLL: Any participant experiencing progression of aPAP lung disease (defined as the disease progression resulting in respiratory failure (PaO2 at rest <60 mmHg of PaO2 > 60 mmHg at rest AND desaturation <90% at rest OR decline in SpO2 of 5% or more during exercise testing) will receive unscheduled rescue WLL.
  Interventions: Procedure: Baseline WLL; Drug: Sargramostim; Procedure: Rescue WLL
- Control Group (Other): Scheduled Baseline WLL: All participants will receive a scheduled bilateral WLL at baseline (month 0).
  Unscheduled Rescue WLL: Any participant experiencing progression of aPAP lung disease (defined as the disease progression resulting in respiratory failure (defined by a resting PaO2 <60 mmHg or > 60 mmHg and desaturation <90% at rest or decline in SpO2 of 5% or more during exercise testing) will receive unscheduled rescue WLL.
  Interventions: Procedure: Baseline WLL; Procedure: Rescue WLL

INTERVENTIONS:
Procedure: Baseline WLL — Scheduled bilateral WLL
Drug: Sargramostim — Inhaled GM-CSF
  Other Names: Leukine®, recombinant granulocyte/macrophage-colony stimulating factor
  Arms: GM-CSF Group
Procedure: Rescue WLL — Unscheduled bilateral WLL

SUMMARY:
This is a prospective, randomized, open-label, long-term, phase 2 study of inhaled granulocyte/macrophage-colony stimulating factor following whole lung lavage therapy in patients with autoimmune pulmonary alveolar proteinosis.

DETAILED DESCRIPTION:
Autoimmune pulmonary alveolar proteinosis (aPAP) is a rare disorder of progressive surfactant accumulation and resulting hypoxemic respiratory failure caused by disruption of granulocyte/macrophage-colony stimulating factor (GM-CSF) signaling, which alveolar macrophages require to remove pulmonary surfactant.

The current therapy of aPAP, whole lung lavage (WLL), is a procedure requiring general anesthesia, endotracheal intubation to isolate each lung, and mechanical ventilation of the untreated lung while the treated lung repeatedly filled with saline and drained while percussing the chest to loosen and emulsify the surfactant and saline to physically remove the excess surfactant.

Inhaled GM-CSF is a promising pharmacotherapeutic approach shown in case reports, small series, moderate open-label studies, and two randomized, double-blinded, placebo-controlled trials to be safe and improve the clinical, physiological, radiological, and biochemical disease manifestations in patients with mild-moderate aPAP. In contrast to the present study, prior studies were too short in duration to permit an evaluation on the requirement for WLL, which aPAP patients require a mean of every 15 months. The present study addressed the effects on WLL by studying patients with moderate-severe aPAP and by utilizing a long-term follow up period.

The study design included a screening visit (month -3) to establish eligibility, an observation period (-3 to 0 months) to establish the presence of progressive/unremitting aPAP and establish disease severity, a pre-WLL visit (-1 month), a baseline visit (month 0) during which all patients received a scheduled, baseline, bilateral WLL, a 10-month, open-label treatment period, and a 20-month follow-up period. Study visits were scheduled at months -3, -1, 0, 1, 3, 6, 10, 18, and 30 months. Patients were randomized by the statistician to the GM-CSF Group (n=9) or the Control Group (n=9). Investigators were blinded to group assignment until after the participant's baseline visit.

Patients randomized to the GM-CSF group (n=9) received inhaled GM-CSF (sargramostim (Leukine®), 250 mcg daily every other week for 12 weeks beginning 1 week after the baseline WLL - termed GM-CSF induction therapy period, followed by a 4-week washout period during which no GM-CSF was administered), and then received inhaled GM-CSF (sargramostim, 250 mcg/day on days 1 and 3 of every 14-day period for 6 months - termed GM-CSF maintenance therapy period). Inhaled GM-CSF (Leukine®) was administered using AKITA2 APIXNEB nebulizer system (Activaero, Vectura GmbH, Germany). Patients randomized to the Control Group (n=9) received no further scheduled treatment. Any patient in either group experiencing with disease progression resulting in respiratory failure (defined as peripheral artery oxygen concentration (PaO2) <60 mmHg at rest or PaO2 >60 mmHg at rest AND a peripheral blood oxygen saturation (SpO2) < 90% OR a decline in SpO2 of 5% or more during exercise), received (unscheduled) rescue WLL and were considered to have failed their assigned intervention (GM-CSF or Control).

The primary outcome measure was time, in months, between the scheduled baseline WLL and first administration of unscheduled 'rescue' WLL (termed 'time to rescue WLL'). Key secondary outcome measures included the response in peripheral arterial oxygen concentration (PaO2), alveolar-arterial difference in oxygen concentration (A-aDO2), diffusing capacity of the lungs for carbon monoxide (DLco), vital capacity, ground glass opacification (GGO) of the lungs measured by visual scoring of chest computed tomography (CT) scans, and serum biomarkers of PAP (carcinoembryonic antigen, Krebs von-Lungren antigen, Cyfra-21.1). Other outcome measures included the Medical Outcomes Study 36-Item Short-Form Health Survey (SF-36), serum GM-CSF autoantibody concentration, the peripheral white blood cell and platelet counts.

The occurrence and timing of rescue WLL administration in each group was evaluated using Kaplan-Meyer analysis. The primary end point was analyzed as the difference in median time to rescue WLL between the GM-CSF group and the Control group. Categorical outcomes were compared using Fisher's exact test. Key secondary end points were evaluated using repeated measures analysis of variance (RM-ANOVA) after adjustment for baseline values, gender, age, and the number of patients at risk at each time point. Secondary outcome measures were also evaluated by comparing the between-group mean (or median) values at each visit using Student's t-test (or Mann-Whitney test) after imputation of missing data using a last observation carried forward approach to reduce selection-type bias by comparing the corresponding group means or medians. All reported p values are two-sided and have not been adjusted for multiple testing. P values of less than 0.05 were considered to indicate statistical significance. Analysis of the primary and key secondary outcomes was performed with the use of Stata software version 14.2. Analyses of secondary outcome measures were performed with the use of Prism for Mac OS software, version 9.51.

Anticipated results were intended to compare the effects of inhaled GM-CSF following baseline WLL to those of baseline WLL alone in patients with moderate to severe aPAP.

ELIGIBILITY:
Inclusion Criteria:

* Female of male 18 years of age or older
* Diagnosis of autoimmune PAP
* Able and willing to provide written informed consent
* Eligible for whole lung lavage determined as the presence of persistent or progressive respiratory failure (PaO2 at rest < 60 mm Hg) or desaturation < 90% or > 5 percentage points during standard exercise

Exclusion Criteria:

* Diagnosis with secondary PAP, congenital PAP, or hereditary PAP
* Contraindication to whole lung lavage
* Contraindication to administration of inhaled GM-CSF
* Chronic lung disease associated with already existing respiratory failure, such as emphysema or pulmonary fibrosis, chronic heart failure, ischemic heart disease, active pulmonary embolism, progressive cancer, and other severe metabolic conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2009-07 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francesca Mariani, MD, Principal Investigator — Fondazione IRCCS Policlinico San Matteo
Locations (1):
- Fondazione IRCCS Policlinico San Matteo, Pavia, PV, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Trapnell BC, Whitsett JA, Nakata K. Pulmonary alveolar proteinosis. N Engl J Med. 2003 Dec 25;349(26):2527-39. doi: 10.1056/NEJMra023226. No abstract available. PMID 14695413
- [Background] Beccaria M, Luisetti M, Rodi G, Corsico A, Zoia MC, Colato S, Pochetti P, Braschi A, Pozzi E, Cerveri I. Long-term durable benefit after whole lung lavage in pulmonary alveolar proteinosis. Eur Respir J. 2004 Apr;23(4):526-31. doi: 10.1183/09031936.04.00102704. PMID 15083749
- [Background] Wylam ME, Ten R, Prakash UB, Nadrous HF, Clawson ML, Anderson PM. Aerosol granulocyte-macrophage colony-stimulating factor for pulmonary alveolar proteinosis. Eur Respir J. 2006 Mar;27(3):585-93. doi: 10.1183/09031936.06.00058305. PMID 16507860
- [Background] Trapnell BC, Inoue Y, Bonella F, Morgan C, Jouneau S, Bendstrup E, Campo I, Papiris SA, Yamaguchi E, Cetinkaya E, Ilkovich MM, Kramer MR, Veltkamp M, Kreuter M, Baba T, Ganslandt C, Tarnow I, Waterer G, Jouhikainen T; IMPALA Trial Investigators. Inhaled Molgramostim Therapy in Autoimmune Pulmonary Alveolar Proteinosis. N Engl J Med. 2020 Oct 22;383(17):1635-1644. doi: 10.1056/NEJMoa1913590. Epub 2020 Sep 7. PMID 32897035
- [Background] Tazawa R, Ueda T, Abe M, Tatsumi K, Eda R, Kondoh S, Morimoto K, Tanaka T, Yamaguchi E, Takahashi A, Oda M, Ishii H, Izumi S, Sugiyama H, Nakagawa A, Tomii K, Suzuki M, Konno S, Ohkouchi S, Tode N, Handa T, Hirai T, Inoue Y, Arai T, Asakawa K, Sakagami T, Hashimoto A, Tanaka T, Takada T, Mikami A, Kitamura N, Nakata K. Inhaled GM-CSF for Pulmonary Alveolar Proteinosis. N Engl J Med. 2019 Sep 5;381(10):923-932. doi: 10.1056/NEJMoa1816216. PMID 31483963

RESULTS

PARTICIPANT FLOW:
Groups:
- Control Group: All participants received a scheduled bilateral whole lung lavage (WLL) at baseline (month 0). Unscheduled rescue WLL was administered, as required, to any participant who experienced progression of pulmonary alveolar proteinosis (PAP) lung disease as defined in the protocol.
- GM-CSF Group: All participants received a scheduled bilateral WLL at baseline (month 0). All participants received inhaled granulocyte/macrophage-colony stimulating factor (GM-CSF) (sargramostim, 250 mcg) administered once daily every other week for 12 consecutive weeks, followed by a 4-week washout period without GM-CSF administration, followed by GM-CSF administration on days 1 and 3 of every consecutive 14-day period for 6 months. Unscheduled rescue WLL was administered, as required, to any participant who experienced progression of PAP lung disease as defined in the protocol.
Period: Overall Study
Arm/Group | Control Group | GM-CSF Group
Started | 9 | 9
Completed | 8 | 8
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- GM-CSF Group: All participants received a scheduled bilateral WLL at baseline (month 0). All participants received inhaled granulocyte/macrophage-colony stimulating factor (GM-CSF) (Sargramostim, 250 mcg) administered once daily every other week for 12 consecutive weeks, followed by a 4-week washout period without administration, followed by administration on days 1 and 3 of every consecutive 14-day period for 6 months. Unscheduled rescue WLL was administered, as required, to any participant who experienced progression of PAP lung disease as defined in the protocol.
- Total: Total of all reporting groups
Arm/Group | Control Group | GM-CSF Group | Total
Number analyzed (Participants) | 9 | 9 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 9 | 18
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 48 (9.2) | 36 (13) | 42 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 5 | 6 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 8 | 9 | 17
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Italy | 9 | 9 | 18

OUTCOME MEASURES:

1. Primary Outcome: Time to Rescue WLL
Description: Time (in months) between the scheduled baseline WLL (at Study Month 0) and the first administration of an unscheduled rescue WLL (during the 30-months after Study Month 0)
Time Frame: 30 months
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Control Group | GM-CSF Group
Number analyzed (Participants) | 9 | 9
Months | 18 [6 to 27] | 30 [30 to 30]
Statistical Analysis 1: Comparison: Control Group vs GM-CSF Group; Test type: Superiority; p = 0.0078, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 12 — Calculated as the median time to rescue WLL in the GM-CSF Group minus the median the time to rescue WLL in the Control Group

2. Secondary Outcome: Number of Patients Requiring a Rescue WLL
Description: Number of patients requiring an unscheduled rescue WLL during the 30-months immediately following administration of the scheduled baseline WLL therapy at Study Month 0.
Time Frame: 30 months
Measure: Number; unit: participants
Arm/Group | Control Group | GM-CSF Group
Number analyzed (Participants) | 9 | 9
participants | 7 | 1
Statistical Analysis 1: Comparison: Control Group vs GM-CSF Group; Test type: Superiority; p = 0.0152, Fisher Exact; Risk Ratio (RR) = 7, 95% CI 2-sided [1.60 to 39.9] — Calculated as risk ratio of rescue WLL in the Control Group compared to the risk ratio of rescue WLL in the GM-CSF Group

3. Secondary Outcome: Between-Group Difference in Mean Partial Pressure of Oxygen (PaO2)
Description: Primary Analysis: Between-group difference in mean PaO2 at each study visit after the scheduled baseline WLL was evaluated using repeated measures analysis of variance (ANOVA) after adjustment for baseline values, gender, age, and the number of patients at risk at each time point.
  Secondary analysis: Between-group difference in mean PaO2 at each visit after imputation of missing data by the last observation carried forward method.
  For both of the primary and secondary analyses, PaO2 is determined from lab values measured for an arterial blood gas procedure.
Time Frame: 30 months
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Control Group | GM-CSF Group
Number analyzed (Participants) | 9 | 9
mmHg
  Pre-WLL ( Month -1) | 51 (12) | 66 (14)
  Baseline (Month 0) | 72 (15) | 82 (11)
  1 month | 70 (14) | 88 (8.4)
  3 months | 68 (10) | 89 (9.2)
  6 months | 73 (11) | 92 (14)
  10 months | 73 (13) | 92 (12)
  18 months | 71 (14) | 90 (16)
  30 months | 71 (14) | 82 (14)
Statistical Analysis 1: Comparison: Control Group vs GM-CSF Group; Test type: Superiority; p < 0.0001, Repeated measures ANOVA; Data was evaluated via repeated measures ANOVA after adjustment for baseline values, gender, age, and number of patients at risk at each time point; Mean Difference (Final Values) = 9.5, 95% CI 2-sided [5.7 to 13.3] — Calculated as the between group difference in the mean PaO2 in the GM-CSF Group minus the between group difference in mean PaO2 in the Control Group
Statistical Analysis 2: Comparison: Control Group vs GM-CSF Group; The secondary analysis includes evaluation of the difference in mean PaO2 between groups at the pre-WLL visit after imputation of missing data using a last observation carried forward method; Test type: Superiority; p = 0.0261, t-test, 2 sided; Mean Difference (Final Values) = 15.10, 95% CI 2-sided [2.04 to 28.16], Standard Error of Mean 6.16 — Calculated as the difference at the pre-WLL visit in the mean PaO2 in the GM-CSF Group minus the mean PaO2 in the Control Group
Statistical Analysis 3: Comparison: Control Group vs GM-CSF Group; The secondary analysis includes evaluation of the difference in mean PaO2 between groups at the baseline visit after imputation of missing data using a last observation carried forward method; Test type: Superiority; p = 0.1521, t-test, 2 sided; Mean Difference (Final Values) = 9.56, 95% CI 2-sided [3.92 to 23.03], Standard Error of Mean 6.36 — Calculated as the difference at the baseline visit in the mean PaO2 in the GM-CSF Group minus the mean PaO2 in the Control Group
Statistical Analysis 4: Comparison: Control Group vs GM-CSF Group; The secondary analysis includes evaluation of the difference in mean PaO2 between groups at the 1-month visit after imputation of missing data using a last observation carried forward method; Test type: Superiority; p = 0.0051, t-test, 2 sided; Mean Difference (Final Values) = 18.04, 95% CI 2-sided [6.26 to 29.82], Standard Error of Mean 5.56 — Calculated as the difference at the 1-month visit in the mean PaO2 in the GM-CSF Group minus the mean PaO2 in the Control Group
Statistical Analysis 5: Comparison: Control Group vs GM-CSF Group; The secondary analysis includes evaluation of the difference in mean PaO2 between groups at the 3-month visit after imputation of missing data using a last observation carried forward method; Test type: Superiority; p = 0.0004, t-test, 2 sided; Mean Difference (Final Values) = 20.26, 95% CI 2-sided [10.63 to 29.88], Standard Error of Mean 4.54 — Calculated as the difference at the 3-month visit in the mean PaO2 in the GM-CSF Group minus the mean PaO2 in the Control Group
Statistical Analysis 6: Comparison: Control Group vs GM-CSF Group; The secondary analysis includes evaluation of the difference in mean PaO2 between groups at the 6-month visit after imputation of missing data using a last observation carried forward method; Test type: Superiority; p = 0.0038, t-test, 2 sided; Mean Difference (Final Values) = 19.91, 95% CI 2-sided [7.43 to 32.40], Standard Error of Mean 5.89 — Calculated as the difference at the 6-month visit in the mean PaO2 in the GM-CSF Group minus the mean PaO2 in the Control Group
Statistical Analysis 7: Comparison: Control Group vs GM-CSF Group; The secondary analysis includes evaluation of the difference in mean PaO2 between groups at the 10-month visit after imputation of missing data using a last observation carried forward method; Test type: Superiority; p = 0.0149, t-test, 2 sided; Mean Difference (Final Values) = 16.92, 95% CI 2-sided [3.81 to 30.03], Standard Error of Mean 6.15 — Calculated as the difference at the 10-month visit in the mean PaO2 in the GM-CSF Group minus the mean PaO2 in the Control Group
Statistical Analysis 8: Comparison: Control Group vs GM-CSF Group; The secondary analysis includes evaluation of the difference in mean PaO2 between groups at the 18-month visit after imputation of missing data using a last observation carried forward method; Test type: Superiority; p = 0.0148, t-test, 2 sided; Mean Difference (Final Values) = 19.02, 95% CI 2-sided [4.26 to 33.79], Standard Error of Mean 6.97 — Calculated as the difference at the 18-month visit in the mean PaO2 in the GM-CSF Group minus the mean PaO2 in the Control Group
Statistical Analysis 9: Comparison: Control Group vs GM-CSF Group; The secondary analysis includes evaluation of the difference in mean PaO2 between groups at the 30-month visit after imputation of missing data using a last observation carried forward method; Test type: Superiority; p = 0.1158, t-test, 2 sided; Mean Difference (Final Values) = 11.00, 95% CI 2-sided [-3.02 to 25.02], Standard Error of Mean 6.62; Calculated as the difference at the 30-month visit in the mean PaO2 in the GM-CSF Group minus the mean PaO2 in the Control Group

4. Secondary Outcome: Between-Group Difference in Mean Alveolar-arterial Difference in Oxygen Concentration (A-aDO2)
Description: Primary Analysis: Between-group difference in mean A-aDO2 at each study visit after the scheduled baseline WLL was evaluated using repeated measures analysis of variance (ANOVA) after adjustment for baseline values, gender, age, and the number of patients at risk at each time point.
  Secondary analysis: Between-group difference in mean A-aDO2 at each visit after imputation of missing data by the last-value carried forward method.
  For both of the primary and secondary analyses, A-aDO2 is calculated from lab values measured for an arterial blood gas, the ambient atmosphere pressure, and fraction of inspired oxygen at the time of the arterial blood gas procedure.
Time Frame: 30 months
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Control Group | GM-CSF Group
Number analyzed (Participants) | 9 | 9
mmHg
  Pre-WLL (Month -1) | 55 (11) | 43 (14)
  Baseline (Month 0) | 33 (15) | 26 (12)
  1 month | 37 (17) | 20 (7.2)
  3 months | 37 (12) | 18 (8.1)
  6 months | 35 (12) | 15 (12)
  10 months | 34 (13) | 18 (12)
  18 months | 35 (13) | 18 (13)
  30 months | 35 (13) | 24 (13)
Statistical Analysis 1: Comparison: Control Group vs GM-CSF Group; Primary analysis; Test type: Superiority; p < 0.0001, Repeated measures ANOVA; [statistical method as in outcome 3, analysis 1]; Mean Difference (Final Values) = -10.1, 95% CI 2-sided [-14.8 to -5.4] — Calculated as the between group difference in the mean value of A-aDO2 in the GM-CSF Group minus the mean value of A-aDO2 in the Control Group
Statistical Analysis 2: Comparison: Control Group vs GM-CSF Group; The secondary analysis includes evaluation of the difference in mean A-aDO2 between groups at the pre-WLL visit after imputation of missing data using a last observation carried forward method; Test type: Superiority; p = 0.0545, t-test, 2 sided; Mean Difference (Final Values) = -12.46, 95% CI 2-sided [-25.19 to 0.27], Standard Error of Mean 6.00 — Calculated as the difference at the pre-WLL visit in the mean A-aDO2 in the GM-CSF Group minus the mean A-aDO2 in the Control Group
Statistical Analysis 3: Comparison: Control Group vs GM-CSF Group; The secondary analysis includes evaluation of the difference in mean A-aDO2 between groups at the baseline visit after imputation of missing data using a last observation carried forward method; Test type: Superiority; p = 0.2802, t-test, 2 sided; Mean Difference (Final Values) = -7.08, 95% CI 2-sided [-20.52 to 6.35], Standard Error of Mean 6.34 — Calculated as the difference at the baseline visit in the mean A-aDO2 in the GM-CSF Group minus the mean A-aDO2 in the Control Group
Statistical Analysis 4: Comparison: Control Group vs GM-CSF Group; The secondary analysis includes evaluation of the difference in mean A-aDO2 between groups at the 1-month visit after imputation of missing data using a last observation carried forward method; Test type: Superiority; p = 0.0148, t-test, 2 sided; Mean Difference (Final Values) = -16.81, 95% CI 2-sided [-29.85 to -3.76], Standard Error of Mean 6.16 — Calculated as the difference at the 1-month visit in the mean A-aDO2 in the GM-CSF Group minus the mean A-aDO2 in the Control Group
Statistical Analysis 5: Comparison: Control Group vs GM-CSF Group; The secondary analysis includes evaluation of the difference in mean A-aDO2 between groups at the 3 -month visit after imputation of missing data using a last observation carried forward method; Test type: Superiority; p = 0.0015, t-test, 2 sided; Mean Difference (Final Values) = -18.77, 95% CI 2-sided [-29.18 to -8.36], Standard Error of Mean 4.91 — Calculated as the difference at the 3-month visit in the mean A-aDO2 in the GM-CSF Group minus the mean A-aDO2 in the Control Group
Statistical Analysis 6: Comparison: Control Group vs GM-CSF Group; The secondary analysis includes evaluation of the difference in mean A-aDO2 between groups at the 6-month visit after imputation of missing data using a last observation carried forward method; Test type: Superiority; p = 0.0049, t-test, 2 sided; Mean Difference (Final Values) = -19.09, 95% CI 2-sided [-31.49 to -6.70], Standard Error of Mean 5.85 — Calculated as the difference at the 6-month visit in the mean A-aDO2 in the GM-CSF Group minus the mean A-aDO2 in the Control Group
Statistical Analysis 7: Comparison: Control Group vs GM-CSF Group; The secondary analysis includes evaluation of the difference in mean A-aDO2 between groups at the 10-month visit after imputation of missing data using a last observation carried forward method; Test type: Superiority; p = 0.0152, t-test, 2 sided; Mean Difference (Final Values) = -15.85, 95% CI 2-sided [-28.23 to -3.48], Standard Error of Mean 5.84 — Calculated as the difference at the 10-month visit in the mean A-aDO2 in the GM-CSF Group minus the mean A-aDO2 in the Control Group
Statistical Analysis 8: Comparison: Control Group vs GM-CSF Group; The secondary analysis includes evaluation of the difference in mean A-aDO2 between groups at the 18-month visit after imputation of missing data using a last observation carried forward method; Test type: Superiority; p = 0.0154, t-test, 2 sided; Mean Difference (Final Values) = -17.01, 95% CI 2-sided [-30.31 to -3.71], Standard Error of Mean 6.27 — Calculated as the difference at the 18-month visit in the mean A-aDO2 in the GM-CSF Group minus the mean A-aDO2 in the Control Group
Statistical Analysis 9: Comparison: Control Group vs GM-CSF Group; The secondary analysis includes evaluation of the difference in mean A-aDO2 between groups at the 30-month visit after imputation of missing data using a last observation carried forward method; Test type: Superiority; p = 0.0921, t-test, 2 sided; Mean Difference (Final Values) = -11.01, 95% CI 2-sided [-24.05 to 2.02], Standard Error of Mean 6.15 — Calculated as the difference at the 30-month visit in the mean A-aDO2 in the GM-CSF Group minus the mean A-aDO2 in the Control Group

5. Secondary Outcome: Between-Group Difference in Mean Diffusion Capacity of the Lungs for Carbon Monoxide (DLCO)
Description: Primary Analysis: Between-group difference in mean DLCO at each study visit after the scheduled baseline WLL was evaluated using repeated measures analysis of variance (ANOVA) after adjustment for baseline values, gender, age, and the number of patients at risk at each time point.
  Secondary analysis: Between-group difference in mean DLCO at each visit after imputation of missing data by the last observation carried forward method.
  For both of the primary and secondary analyses, DLCO is determined from pulmonary function tests.
Time Frame: 30 months
Measure: Mean (Standard Deviation); unit: % predicted
Arm/Group | Control Group | GM-CSF Group
Number analyzed (Participants) | 9 | 9
% predicted
  Pre-WLL (Month -1) | 38 (14) | 46 (16)
  Baseline (Month 0) | 50 (14) | 55 (14)
  1 Month | 55 (13) | 68 (15)
  3 months | 62 (16) | 72 (17)
  6 months | 58 (20) | 71 (15)
  10 months | 59 (20) | 70 (15)
  18 months | 58 (21) | 71 (17)
  30 months | 59 (21) | 63 (16)
Statistical Analysis 1: Comparison: Control Group vs GM-CSF Group; Primary Analysis; Test type: Superiority; p = 0.0220, Repeated measures ANOVA; [statistical method as in outcome 3, analysis 1]; Mean Difference (Final Values) = 11.6, 95% CI 2-sided [1.9 to 21.3] — Calculated as the between group difference in the mean value of the DLCO in the GM-CSF Group minus the mean value of the DLCO in the Control Group
Statistical Analysis 2: Comparison: Control Group vs GM-CSF Group; The secondary analysis includes evaluation of the difference in mean DLCO between groups at the Pre-WLL visit after imputation of missing data using a last observation carried forward method; Test type: Superiority; p = 0.3186, t-test, 2 sided; Mean Difference (Final Values) = 8.29, 95% CI 2-sided [-9.06 to 25.63], Standard Error of Mean 7.96 — Calculated as the difference at the Pre-WLL visit in the mean DLCO in the GM-CSF Group minus the mean DLCO in the Control Group
Statistical Analysis 3: Comparison: Control Group vs GM-CSF Group; The secondary analysis includes evaluation of the difference in mean DLCO between groups at the baseline visit after imputation of missing data using a last observation carried forward method; Test type: Superiority; p = 0.4111, t-test, 2 sided; Mean Difference (Final Values) = 5.56, 95% CI 2-sided [-8.40 to 19.51], Standard Error of Mean 6.58 — Calculated as the difference at the baseline visit in the mean DLCO in the GM-CSF Group minus the mean DLCO in the Control Group
Statistical Analysis 4: Comparison: Control Group vs GM-CSF Group; The secondary analysis includes evaluation of the difference in mean DLCO between groups at the 1-month visit after imputation of missing data using a last observation carried forward method; Test type: Superiority; p = 0.0658, t-test, 2 sided; Mean Difference (Final Values) = 12.89, 95% CI 2-sided [-0.95 to 26.73], Standard Error of Mean 6.53 — Calculated as the difference at the 1-month visit in the mean DLCO in the GM-CSF Group minus the mean DLCO in the Control Group
Statistical Analysis 5: Comparison: Control Group vs GM-CSF Group; The secondary analysis includes evaluation of the difference in mean DLCO between groups at the 3-month visit after imputation of missing data using a last observation carried forward method; Test type: Superiority; p = 0.2287, t-test, 2 sided; Mean Difference (Final Values) = 9.78, 95% CI 2-sided [-6.78 to 26.34], Standard Error of Mean 7.81 — Calculated as the difference at the 3-month visit in the mean DLCO in the GM-CSF Group minus the mean DLCO in the Control Group
Statistical Analysis 6: Comparison: Control Group vs GM-CSF Group; The secondary analysis includes evaluation of the difference in mean DLCO between groups at the 6-month visit after imputation of missing data using a last observation carried forward method; Test type: Superiority; p = 0.1432, t-test, 2 sided; Mean Difference (Final Values) = 12.86, 95% CI 2-sided [-4.86 to 30.64], Standard Error of Mean 8.37 — Calculated as the difference at the 6-month visit in the mean DLCO in the GM-CSF Group minus the mean DLCO in the Control Group
Statistical Analysis 7: Comparison: Control Group vs GM-CSF Group; The secondary analysis includes evaluation of the difference in mean DLCO between groups at the 10-month visit after imputation of missing data using a last observation carried forward method; Test type: Superiority; p = 0.1833, t-test, 2 sided; Mean Difference (Final Values) = 11.78, 95% CI 2-sided [-6.17 to 29.73], Standard Error of Mean 8.47 — Calculated as the difference at the 10-month visit in the mean DLCO in the GM-CSF Group minus the mean DLCO in the Control Group
Statistical Analysis 8: Comparison: Control Group vs GM-CSF Group; The secondary analysis includes evaluation of the difference in mean DLCO between groups at the 18-month visit after imputation of missing data using a last observation carried forward method; Test type: Superiority; p = 0.1888, t-test, 2 sided; Mean Difference (Final Values) = 12.67, 95% CI 2-sided [-6.90 to 32.23], Standard Error of Mean 9.23 — Calculated as the difference at the 18-month visit in the mean DLCO in the GM-CSF Group minus the mean DLCO in the Control Group
Statistical Analysis 9: Comparison: Control Group vs GM-CSF Group; The secondary analysis includes evaluation of the difference in mean DLCO between groups at the 30-month visit after imputation of missing data using a last observation carried forward method; Test type: Superiority; p = 0.6374, t-test, 2 sided; Mean Difference (Final Values) = 4.22, 95% CI 2-sided [-14.41 to 22.85], Standard Error of Mean 8.79 — Calculated as the difference at the 30-month visit in the mean DLCO in the GM-CSF Group minus the mean DLCO in the Control Group

6. Secondary Outcome: Between-Group Difference in Mean Vital Capacity (VC)
Description: Primary Analysis: Between-group difference in mean VC at each study visit after the scheduled baseline WLL was evaluated using repeated measures analysis of variance (ANOVA) after adjustment for baseline values, gender, age, and the number of patients at risk at each time point.
  Secondary analysis: Between-group difference in mean VC at each visit after imputation of missing data by the last observation carried forward method.
  For both of the primary and secondary analyses, VC is determined from pulmonary function tests.
Time Frame: 30 months
Measure: Mean (Standard Deviation); unit: % predicted
Arm/Group | Control Group | GM-CSF Group
Number analyzed (Participants) | 9 | 9
% predicted
  Pre-WLL (Month -1) | 60 (16) | 64 (13)
  Baseline (Month 0) | 74 (11) | 76 (17)
  1 month | 75 (17) | 76 (16)
  3 months | 78 (17) | 80 (15)
  6 months | 78 (15) | 84 (20)
  10 months | 78 (14) | 82 (18)
  18 months | 78 (13) | 83 (21)
  30 months | 77 (13) | 79 (17)
Statistical Analysis 1: Comparison: Control Group vs GM-CSF Group; Primary Analysis; Test type: Superiority; p = 0.5320, Repeated measures ANOVA; [statistical method as in outcome 3, analysis 1]; Mean Difference (Final Values) = 2.0, 95% CI 2-sided [-5.30 to 9.90] — Calculated as the between group difference in the mean value of VC in the GM-CSF Group minus the mean value of VC in the Control Group
Statistical Analysis 2: Comparison: Control Group vs GM-CSF Group; The secondary analysis includes evaluation of the difference in mean VC between groups at the Pre-WLL visit after imputation of missing data using a last observation carried forward method; Test type: Superiority; p = 0.6772, t-test, 2 sided; Mean Difference (Final Values) = 3.21, 95% CI 2-sided [-13.09 to 19.52], Standard Error of Mean 7.55 — Calculated as the difference at the Pre-WLL visit in the mean VC in the GM-CSF Group minus the mean VC in the Control Group
Statistical Analysis 3: Comparison: Control Group vs GM-CSF Group; The secondary analysis includes evaluation of the difference in mean VC between groups at the baseline visit after imputation of missing data using a last observation carried forward method; Test type: Superiority; p = 0.8320, t-test, 2 sided; Mean Difference (Final Values) = 1.44, 95% CI 2-sided [-12.52 to 15.64], Standard Error of Mean 6.70 — Calculated as the difference at the baseline visit in the mean VC in the GM-CSF Group minus the mean VC in the Control Group
Statistical Analysis 4: Comparison: Control Group vs GM-CSF Group; The secondary analysis includes evaluation of the difference in mean VC between groups at the 1-month visit after imputation of missing data using a last observation carried forward method; Test type: Superiority; p = 0.8532, t-test, 2 sided; Mean Difference (Final Values) = 1.47, 95% CI 2-sided [-15.19 to 18.14], Standard Error of Mean 7.82 — Calculated as the difference at the 1-month visit in the mean VC in the GM-CSF Group minus the mean VC in the Control Group
Statistical Analysis 5: Comparison: Control Group vs GM-CSF Group; The secondary analysis includes evaluation of the difference in mean VC between groups at the 3-month visit after imputation of missing data using a last observation carried forward method; Test type: Superiority; p = 0.7752, t-test, 2 sided; Mean Difference (Final Values) = 2.22, 95% CI 2-sided [-14.00 to 18.44], Standard Error of Mean 7.66 — Calculated as the difference at the 3-month visit in the mean VC in the GM-CSF Group minus the mean VC in the Control Group
Statistical Analysis 6: Comparison: Control Group vs GM-CSF Group; The secondary analysis includes evaluation of the difference in mean VC between groups at the 6-month visit after imputation of missing data using a last observation carried forward method; Test type: Superiority; p = 0.5174, t-test, 2 sided; Mean Difference (Final Values) = 5.74, 95% CI 2-sided [-12.70 to 24.18], Standard Error of Mean 8.65 — Calculated as the difference at the 6-month visit in the mean value of VC in the GM-CSF Group minus the mean value of VC in the Control Group
Statistical Analysis 7: Comparison: Control Group vs GM-CSF Group; The secondary analysis includes evaluation of the difference in mean VC between groups at the 10-month visit after imputation of missing data using a last observation carried forward method; Test type: Superiority; p = 0.6393, t-test, 2 sided; Mean Difference (Final Values) = 3.67, 95% CI 2-sided [-12.61 to 19.94], Standard Error of Mean 7.68 — Calculated as the difference at the 10-month visit in the mean VC in the GM-CSF Group minus the mean VC in the Control Group
Statistical Analysis 8: Comparison: Control Group vs GM-CSF Group; The secondary analysis includes evaluation of the difference in mean VC between groups at the 18-month visit after imputation of missing data using a last observation carried forward method; Test type: Superiority; p = 0.5361, t-test, 2 sided; Mean Difference (Final Values) = 5.22, 95% CI 2-sided [-12.28 to 22.73], Standard Error of Mean 8.26 — Calculated as the difference at the 18-month visit in the mean VC in the GM-CSF Group minus the mean VC in the Control Group
Statistical Analysis 9: Comparison: Control Group vs GM-CSF Group; The secondary analysis includes evaluation of the difference in mean VC between groups at the 30-month visit after imputation of missing data using a last observation carried forward method; Test type: Superiority; p = 0.8159, t-test, 2 sided; Mean Difference (Final Values) = 1.67, 95% CI 2-sided [-13.26 to 16.60], Standard Error of Mean 7.04; Calculated as the difference at the 30-month visit in the mean VC in the GM-CSF Group minus the mean VC in the Control Group

7. Secondary Outcome: Between-Group Difference in Mean Chest Computed Tomography Ground Glass Opacification (GGO) Score
Description: Primary Analysis: Between-group difference in median GGO Score at each study visit after the scheduled baseline WLL was evaluated using repeated measures analysis of variance (ANOVA) after adjustment for baseline values, gender, age, and the number of patients at risk at each time point.
  Secondary analysis: Between-group difference in median GGO Score at each visit after imputation of missing data by the last observation carried forward method.
  For both of the primary and secondary analyses, the degree of severity of lung disease was calculated by determining the number of segments affected. The following scale was used:
  Grade 1 = 1 segment affected Grade 2 = 2 - 5 segments affected Grade 3 = 6 - 9 segments affected Grade 4 = 10 - 14 segments affected Grade 5 = > 14 affected segments
Time Frame: 30 months
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Control Group | GM-CSF Group
Number analyzed (Participants) | 9 | 9
score on a scale
  Pre-WLL (Month -1) | 5 [5 to 5] | 5 [5 to 5]
  3 months | 4 [4 to 5] | 3 [2 to 4]
  10 months | 4 [4 to 5] | 3 [2 to 4]
  18 months | 4 [4 to 5] | 3 [2 to 4]
  30 months | 4 [4 to 5] | 4 [3 to 5]
Statistical Analysis 1: Comparison: Control Group vs GM-CSF Group; Primary Analysis; Test type: Superiority; p = 0.0530, Repeated measures ANOVA; [statistical method as in outcome 3, analysis 1]; Mean Difference (Final Values) = -0.822, 95% CI 2-sided [-1.70 to 0.01] — Calculated as the between group difference in the median value of the GGO Score in the GM-CSF Group minus the median value of the GGO Score in the Control Group
Statistical Analysis 2: Comparison: Control Group; The secondary analysis includes evaluation of the difference in median GGO Score between groups at the Pre-WLL visit after imputation of missing data using a last observation carried forward method; Test type: Superiority; p > 0.9999, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 0.00 — Calculated as the difference at the Pre-WLL visit in the median GGO Score in the GM-CSF Group minus the median GGO Score in the Control Group
Statistical Analysis 3: Comparison: Control Group vs GM-CSF Group; The secondary analysis includes evaluation of the difference in median GGO Score between groups at the 3-month visit after imputation of missing data using a last observation carried forward method; Test type: Superiority; p = 0.0332, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = -1.00 — Calculated as the difference at the 3-month visit in the median GGO Score in the GM-CSF Group minus the median GGO Score in the Control Group
Statistical Analysis 4: Comparison: Control Group vs GM-CSF Group; The secondary analysis includes evaluation of the difference in median GGO Score between groups at the 10-month visit after imputation of missing data using a last observation carried forward method; Test type: Superiority; p = 0.0676, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = -1.00 — Calculated as the difference at the 10-month visit in the median GGO Score in the GM-CSF Group minus the median GGO Score in the Control Group
Statistical Analysis 5: Comparison: Control Group vs GM-CSF Group; The secondary analysis includes evaluation of the difference in median GGO Score between groups at the 18-month visit after imputation of missing data using a last observation carried forward method; Test type: Superiority; p = 0.0629, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = -1.00 — Calculated as the difference at the 18-month visit in the median GGO Score in the GM-CSF Group minus the median GGO Score in the Control Group
Statistical Analysis 6: Comparison: Control Group vs GM-CSF Group; The secondary analysis includes evaluation of the difference in median GGO Score between groups at the 30-month visit after imputation of missing data using a last observation carried forward method; Test type: Superiority; p > 0.9999, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 0.00 — Calculated as the difference at the 30-month visit in the median GGO Score in the GM-CSF Group minus the median GGO Score in the Control Group

8. Secondary Outcome: Between-Group Difference in Median Serum Carcinoembryonic Antigen (CEA) Levels
Description: Primary Analysis: Between-group difference in median serum CEA levels at each study visit after the scheduled baseline WLL was evaluated using repeated measures analysis of variance (ANOVA) after adjustment for baseline values, gender, age, and the number of patients at risk at each time point.
  Secondary analysis: Between-group difference in serum CEA levels at each visit after imputation of missing data by the last observation carried forward method.
  For both of the primary and secondary analyses, the serum CEA levels were determined via enzyme linked immunosorbent assay (ELISA).
Time Frame: 30 months
Measure: Median (Inter-Quartile Range); unit: ng/ml
Arm/Group | Control Group | GM-CSF Group
Number analyzed (Participants) | 9 | 9
ng/ml
  Pre-WLL (Month -1) | 18 [10 to 41] | 6 [4 to 12]
  Baseline (Month 0) | 8 [7 to 17] | 5 [3 to 9]
  1 month | 6 [5 to 21] | 3 [2 to 5]
  3 months | 8 [4 to 22] | 4 [2 to 5]
  6 months | 10 [4 to 21] | 3 [2 to 3]
  10 months | 9 [4 to 21] | 2 [2 to 3]
  18 months | 9 [5 to 19] | 3 [2 to 4]
  30 months | 8 [5 to 19] | 5 [3 to 5]
Statistical Analysis 1: Comparison: Control Group vs GM-CSF Group; Primary Analysis; Test type: Superiority; p = 0.0010, Repeated measures ANOVA; [statistical method as in outcome 3, analysis 1]; Mean Difference (Final Values) = -0.47, 95% CI 2-sided [-0.71 to -0.22] — Calculated as the between group difference in the CEA levels in the GM-CSF Group minus the CEA levels in the Control Group
Statistical Analysis 2: Comparison: Control Group vs GM-CSF Group; The secondary analysis includes evaluation of the difference in median serum CEA levels between groups at the Pre-WLL visit after imputation of missing data using a last observation carried forward method; Test type: Superiority; p = 0.0059, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = -12 — Calculated as the difference at the Pre-WLL visit in the median serum CEA levels in the GM-CSF Group minus the median serum CEA levels in the Control Group
Statistical Analysis 3: Comparison: Control Group vs GM-CSF Group; The secondary analysis includes evaluation of the difference in median serum CEA levels between groups at the baseline visit after imputation of missing data using a last observation carried forward method; Test type: Superiority; p = 0.0382, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = -3.45 — Calculated as the difference at the baseline visit in the median serum CEA levels in the GM-CSF Group minus the median serum CEA levels in the Control Group
Statistical Analysis 4: Comparison: Control Group vs GM-CSF Group; The secondary analysis includes evaluation of the difference in median serum CEA levels between groups at the 1-month visit after imputation of missing data using a last observation carried forward method; Test type: Superiority; p = 0.0770, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = -3.20 — Calculated as the difference at the 1-month visit in the median serum CEA levels in the GM-CSF Group minus the median serum CEA levels in the Control Group
Statistical Analysis 5: Comparison: Control Group vs GM-CSF Group; The secondary analysis includes evaluation of the difference in median serum CEA levels between groups at the 3-month visit after imputation of missing data using a last observation carried forward method; Test type: Superiority; p = 0.0400, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = -4.00 — Calculated as the difference at the 3-month visit in the median serum CEA levels in the GM-CSF Group minus the median serum CEA levels in the Control Group
Statistical Analysis 6: Comparison: Control Group vs GM-CSF Group; The secondary analysis includes evaluation of the difference in median serum CEA levels between groups at the 6-month visit after imputation of missing data using a last observation carried forward method; Test type: Superiority; p = 0.0142, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = -7.90 — Calculated as the difference at the 6-month visit in the median serum CEA levels in the GM-CSF Group minus the median serum CEA levels in the Control Group
Statistical Analysis 7: Comparison: Control Group vs GM-CSF Group; The secondary analysis includes evaluation of the difference in median serum CEA levels between groups at the 10-month visit after imputation of missing data using a last observation carried forward method; Test type: Superiority; p = 0.0071, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = -6.50 — Calculated as the difference at the 10-month visit in the median serum CEA levels in the GM-CSF Group minus the median serum CEA levels in the Control Group
Statistical Analysis 8: Comparison: Control Group vs GM-CSF Group; The secondary analysis includes evaluation of the difference in median serum CEA levels between groups at the 18-month visit after imputation of missing data using a last observation carried forward method; Test type: Superiority; p = 0.0137, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = -5.60 — Calculated as the difference at the 18-month visit in the median serum CEA levels in the GM-CSF Group minus the median serum CEA levels in the Control Group
Statistical Analysis 9: Comparison: Control Group vs GM-CSF Group; The secondary analysis includes evaluation of the difference in median serum CEA levels between groups at the 30-month visit after imputation of missing data using a last observation carried forward method; Test type: Superiority; p = 0.0315, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = -3.20 — Calculated as the difference at the 30-month visit in the median serum CEA levels in the GM-CSF Group minus the median serum CEA levels in the Control Group

9. Secondary Outcome: Between-Group Difference in Mean Serum Krebs Von-Lungren 6 Antigen (KL-6) Levels
Description: Primary Analysis: Between-group difference in median serum KL-6 levels at each study visit after the scheduled baseline WLL was evaluated using repeated measures analysis of variance (ANOVA) after adjustment for baseline values, gender, age, and the number of patients at risk at each time point.
  Secondary analysis: Between-group difference in serum KL-6 levels at each visit after imputation of missing data by the last observation carried forward method.
  For both of the primary and secondary analyses, the serum KL-6 levels were determined via enzyme linked immunosorbent assay (ELISA).
Time Frame: 30 months
Measure: Median (Inter-Quartile Range); unit: U/ml
Arm/Group | Control Group | GM-CSF Group
Number analyzed (Participants) | 9 | 9
U/ml
  Pre-WLL (Month -1) | 9023 [6660 to 19205] | 5758 [3247 to 7759]
  Baseline (Month 0) | 10556 [6501 to 18734] | 5538 [1738 to 7287]
  1 month | 8744 [6340 to 14413] | 2401 [1348 to 14828]
  3 months | 6524 [2296 to 18562] | 2422 [718 to 11473]
  6 months | 8934 [808 to 13494] | 2117 [648 to 29300]
  10 months | 8116 [712 to 14141] | 6546 [1218 to 13697]
  18 months | 7314 [1714 to 11335] | 3114 [1330 to 5742]
  30 months | 5755 [1714 to 8257] | 1448 [666 to 8539]
Statistical Analysis 1: Comparison: Control Group vs GM-CSF Group; Primary Analysis; Test type: Superiority; p = 0.0300, Repeated measures ANOVA; [statistical method as in outcome 3, analysis 1]; Mean Difference (Final Values) = -3689, 95% CI 2-sided [-6972 to -406] — Calculated as the between group difference in the KL-6 levels in the GM-CSF Group minus the KL-6 levels in the Control Group
Statistical Analysis 2: Comparison: Control Group vs GM-CSF Group; The secondary analysis includes evaluation of the difference in median serum KL-6 levels between groups at the Pre-WLL visit after imputation of missing data using a last observation carried forward method; Test type: Superiority; p = 0.0770, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = -3265 — Calculated as the difference at the Pre-WLL visit in the median serum KL-6 levels in the GM-CSF Group minus the median KL-6 levels in the Control Group
Statistical Analysis 3: Comparison: Control Group vs GM-CSF Group; The secondary analysis includes evaluation of the difference in median serum KL-6 levels between groups at the baseline visit after imputation of missing data using a last observation carried forward method; Test type: Superiority; p = 0.0745, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = -5018 — Calculated as the difference at the baseline visit in the median serum KL-6 levels in the GM-CSF Group minus the median KL-6 levels in the Control Group
Statistical Analysis 4: Comparison: Control Group vs GM-CSF Group; The secondary analysis includes evaluation of the difference in median serum KL-6 levels between groups at the 1-month visit after imputation of missing data using a last observation carried forward method; Test type: Superiority; p = 0.2581, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = -6343 — Calculated as the difference at the 1-month visit in the median serum KL-6 levels in the GM-CSF Group minus the median KL-6 levels in the Control Group
Statistical Analysis 5: Comparison: Control Group vs GM-CSF Group; The secondary analysis includes evaluation of the difference in median serum KL-6 levels between groups at the 3-month visit after imputation of missing data using a last observation carried forward method; Test type: Superiority; p = 0.4894, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = -4102 — Calculated as the difference at the 3-month visit in the median serum KL-6 levels in the GM-CSF Group minus the median KL-6 levels in the Control Group
Statistical Analysis 6: Comparison: Control Group vs GM-CSF Group; The secondary analysis includes evaluation of the difference in median serum KL-6 levels between groups at the 6-month visit after imputation of missing data using a last observation carried forward method; Test type: Superiority; p > 0.9999, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = -6818 — Calculated as the difference at the 6-month visit in the median serum KL-6 levels in the GM-CSF Group minus the median KL-6 levels in the Control Group
Statistical Analysis 7: Comparison: Control Group vs GM-CSF Group; The secondary analysis includes evaluation of the difference in median serum KL-6 levels between groups at the 10-month visit after imputation of missing data using a last observation carried forward method; Test type: Superiority; p = 0.8633, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = -1570 — Calculated as the difference at the 10-month visit in the median serum KL-6 levels in the GM-CSF Group minus the median KL-6 levels in the Control Group
Statistical Analysis 8: Comparison: Control Group vs GM-CSF Group; The secondary analysis includes evaluation of the difference in median serum KL-6 levels between groups at the 18-month visit after imputation of missing data using a last observation carried forward method; Test type: Superiority; p = 0.3401, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = -4200 — Calculated as the difference at the 18-month visit in the median serum KL-6 levels in the GM-CSF Group minus the median KL-6 levels in the Control Group
Statistical Analysis 9: Comparison: Control Group vs GM-CSF Group; The secondary analysis includes evaluation of the difference in median serum KL-6 levels between groups at the 30-month visit after imputation of missing data using a last observation carried forward method; Test type: Superiority; p = 0.2973, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = -4307 — Calculated as the difference at the 30-month visit in the median serum KL-6 levels in the GM-CSF Group minus the median KL-6 levels in the Control Group

10. Secondary Outcome: Between-Group Difference in Mean Serum Cytokeratin-19 Fragment (Cyfra21.1) Levels
Description: Primary Analysis: Between-group difference in mean serum Cyfra21.1 levels at each study visit after the scheduled baseline WLL was evaluated using repeated measures analysis of variance (ANOVA) after adjustment for baseline values, gender, age, and the number of patients at risk at each time point.
  Secondary analysis: Between-group difference in serum Cyfra21.1 levels at each visit after imputation of missing data by the last observation carried forward method.
  For both of the primary and secondary analyses, the serum Cyfra21.1 levels were determined via enzyme linked immunosorbent assay (ELISA).
Time Frame: 30 months
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Control Group | GM-CSF Group
Number analyzed (Participants) | 9 | 9
ng/ml
  Pre-WLL (Month -1) | 27 (17) | 13 (8)
  Baseline (Month 0) | 10 (6) | 6 (2)
  1 month | 11 (7) | 5 (2)
  3 months | 10 (5) | 5 (2)
  6 months | 9 (7) | 4 (2)
  10 months | 9 (6) | 4 (2)
  18 months | 8 (7) | 4 (2)
  30 months | 8 (7) | 5 (2)
Statistical Analysis 1: Comparison: Control Group vs GM-CSF Group; Primary Analysis; Test type: Superiority; p = 0.220, Repeated measures ANOVA; Mean Difference (Final Values) = -0.24, 95% CI 2-sided [-0.44 to -0.04] — Calculated as the between group difference in the serum Cyfra21.1 levels in the GM-CSF Group minus the serum Cyfra21.1 levels in the Control Group
Statistical Analysis 2: Comparison: Control Group vs GM-CSF Group; •The secondary analysis includes evaluation of the difference in mean serum Cyfra21.1 levels between groups at the Pre-WLL visit after imputation of missing data using a last observation carried forward method; Test type: Superiority; p = 0.0560, t-test, 2 sided; Mean Difference (Final Values) = -14.19, 95% CI 2-sided [-28.80 to 0.42], Standard Error of Mean 6.76 — Calculated as the difference at the Pre-WLL visit in the mean serum Cyfra21.1 levels in the GM-CSF Group minus the mean serum Cyfra21.1 levels in the Control Group
Statistical Analysis 3: Comparison: Control Group vs GM-CSF Group; The secondary analysis includes evaluation of the difference in mean serum Cyfra21.1 levels between groups at the baseline visit after imputation of missing data using a last observation carried forward method; Test type: Superiority; p = 0.0648, t-test, 2 sided; Mean Difference (Final Values) = -4.26, 95% CI 2-sided [-8.80 to 0.29], Standard Error of Mean 2.15 — Calculated as the difference at the baseline visit in the mean serum Cyfra21.1 levels in the GM-CSF Group minus the mean serum Cyfra21.1 levels in the Control Group
Statistical Analysis 4: Comparison: Control Group vs GM-CSF Group; The secondary analysis includes evaluation of the difference in mean serum Cyfra21.1 levels between groups at the 1-month visit after imputation of missing data using a last observation carried forward method; Test type: Superiority; p = 0.0175, t-test, 2 sided; Mean Difference (Final Values) = -6.27, 95% CI 2-sided [-11.28 to -1.25], Standard Error of Mean 2.36 — Calculated as the difference at the 1-month visit in the mean serum Cyfra21.1 levels in the GM-CSF Group minus the mean serum Cyfra21.1 levels in the Control Group
Statistical Analysis 5: Comparison: Control Group vs GM-CSF Group; The secondary analysis includes evaluation of the difference in mean serum Cyfra21.1 levels between groups at the 3-month visit after imputation of missing data using a last observation carried forward method; Test type: Superiority; p = 0.0148, t-test, 2 sided; Mean Difference (Final Values) = -16.81, 95% CI 2-sided [-29.85 to -3.76], Standard Error of Mean 6.16 — Calculated as the difference at the 3-month visit in the mean serum Cyfra21.1 levels in the GM-CSF Group minus the mean serum Cyfra21.1 levels in the Control Group
Statistical Analysis 6: Comparison: Control Group vs GM-CSF Group; The secondary analysis includes evaluation of the difference in mean serum Cyfra21.1 levels between groups at the 6-month visit after imputation of missing data using a last observation carried forward method; Test type: Superiority; p = 0.0089, t-test, 2 sided; Mean Difference (Final Values) = -5.41, 95% CI 2-sided [-9.27 to -1.56], Standard Error of Mean 1.82 — Calculated as the difference at the 6-month visit in the mean serum Cyfra21.1 levels in the GM-CSF Group minus the mean serum Cyfra21.1 levels in the Control Group
Statistical Analysis 7: Comparison: Control Group vs GM-CSF Group; The secondary analysis includes evaluation of the difference in mean serum Cyfra21.1 levels between groups at the 10-month visit after imputation of missing data using a last observation carried forward method; Test type: Superiority; p = 0.0343, t-test, 2 sided; Mean Difference (Final Values) = -5.18, 95% CI 2-sided [-9.92 to -0.43], Standard Error of Mean 2.24 — Calculated as the difference at the 10-month visit in the mean serum Cyfra21.1 levels in the GM-CSF Group minus the mean serum Cyfra21.1 levels in the Control Group
Statistical Analysis 8: Comparison: Control Group vs GM-CSF Group; The secondary analysis includes evaluation of the difference in mean serum Cyfra21.1 levels between groups at the 18-month visit after imputation of missing data using a last observation carried forward method; Test type: Superiority; p = 0.0871, t-test, 2 sided; Mean Difference (Final Values) = -4.26, 95% CI 2-sided [-9.21 to 0.69], Standard Error of Mean 2.33 — Calculated as the difference at the 18-month visit in the mean serum Cyfra21.1 levels in the GM-CSF Group minus the mean serum Cyfra21.1 levels in the Control Group
Statistical Analysis 9: Comparison: Control Group vs GM-CSF Group; The secondary analysis includes evaluation of the difference in mean serum Cyfra21.1 levels between groups at the 30-month visit after imputation of missing data using a last observation carried forward method; Test type: Superiority; p = 0.2265, t-test, 2 sided; Mean Difference (Final Values) = -3.01, 95% CI 2-sided [-8.09 to 2.06], Standard Error of Mean 2.40 — Calculated as the difference at the 30-month visit in the mean serum Cyfra21.1 levels in the GM-CSF Group minus the mean serum Cyfra21.1 levels in the Control Group

11. Secondary Outcome: Between-Group Difference in Median Serum GM-CSF Autoantibody (GMAb) Levels
Description: Analysis Method: Between-group difference in serum GMAb levels at each visit after imputation of missing data by the last observation carried forward method.
  The serum GMAb levels were determined via enzyme linked immunosorbent assay (ELISA).
Time Frame: 30 months
Measure: Median (Inter-Quartile Range); unit: mcg/ml
Arm/Group | Control Group | GM-CSF Group
Number analyzed (Participants) | 9 | 9
mcg/ml
  Pre-WLL (Month -1) | 23 [11 to 47] | 32 [18 to 59]
  Baseline (Month 0) | 20 [9 to 27] | 28 [19 to 61]
  1 month | 25 [12 to 48] | 30 [17 to 59]
  3 months | 27 [10 to 47] | 34 [26 to 62]
  6 months | 22 [10 to 54] | 36 [23 to 51]
  10 months | 22 [10 to 51] | 33 [21 to 41]
  18 months | 19 [9 to 50] | 24 [15 to 32]
  30 months | 19 [9 to 50] | 12 [9 to 33]
Statistical Analysis 1: Comparison: Control Group vs GM-CSF Group; The secondary analysis includes evaluation of the difference in median serum GMAb levels between groups at the Pre-WLL visit after imputation of missing data using a last observation carried forward method; Test type: Superiority; p = 0.3865, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 8.78 — Calculated as the difference at the Pre-WLL visit in the median serum GMAb levels in the GM-CSF Group minus the median serum GMAb levels in the Control Group
Statistical Analysis 2: Comparison: Control Group vs GM-CSF Group; The secondary analysis includes evaluation of the difference in median serum GMAb levels between groups at the baseline visit after imputation of missing data using a last observation carried forward method; Test type: Superiority; p = 0.1672, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 7.82 — Calculated as the difference at the baseline visit in the median serum GMAb levels in the GM-CSF Group minus the median serum GMAb levels in the Control Group
Statistical Analysis 3: Comparison: Control Group vs GM-CSF Group; The secondary analysis includes evaluation of the difference in median serum GMAb levels between groups at the 1-month visit after imputation of missing data using a last observation carried forward method; Test type: Superiority; p = 0.4363, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 4.24 — Calculated as the difference at the 1-month visit in the median serum GMAb levels in the GM-CSF Group minus the median serum GMAb levels in the Control Group
Statistical Analysis 4: Comparison: Control Group vs GM-CSF Group; The secondary analysis includes evaluation of the difference in median serum GMAb levels between groups at the 3-month visit after imputation of missing data using a last observation carried forward method; Test type: Superiority; p = 0.1615, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 7.34 — Calculated as the difference at the 3-month visit in the median serum GMAb levels in the GM-CSF Group minus the median serum GMAb levels in the Control Group
Statistical Analysis 5: Comparison: Control Group vs GM-CSF Group; The secondary analysis includes evaluation of the difference in median serum GMAb levels between groups at the 6-month visit after imputation of missing data using a last observation carried forward method; Test type: Superiority; p = 0.1615, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 13.71 — Calculated as the difference at the 6-month visit in the median serum GMAb levels in the GM-CSF Group minus the median serum GMAb levels in the Control Group
Statistical Analysis 6: Comparison: Control Group vs GM-CSF Group; The secondary analysis includes evaluation of the difference in median serum GMAb levels between groups at the 10-month visit after imputation of missing data using a last observation carried forward method; Test type: Superiority; p = 0.3865, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 11.10 — Calculated as the difference at the 10-month visit in the median serum GMAb levels in the GM-CSF Group minus the median serum GMAb levels in the Control Group
Statistical Analysis 7: Comparison: Control Group vs GM-CSF Group; The secondary analysis includes evaluation of the difference in median serum GMAb levels between groups at the 18-month visit after imputation of missing data using a last observation carried forward method; Test type: Superiority; p = 0.6475, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 5.40 — • Calculated as the difference at the 18-month visit in the median serum GMAb levels in the GM-CSF Group minus the median serum GMAb levels in the Control Group
Statistical Analysis 8: Comparison: Control Group vs GM-CSF Group; The secondary analysis includes evaluation of the difference in median serum GMAb levels between groups at the 30-month visit after imputation of missing data using a last observation carried forward method; Test type: Superiority; p = 0.6481, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = -7.00 — Calculated as the difference at the 30-month visit in the median serum GMAb levels in the GM-CSF Group minus the median serum GMAb levels in the Control Group

12. Secondary Outcome: Between-Group Difference in Mean White Blood Cell (WBC) Counts
Description: Analysis Method: Between-group difference in WBC counts at each visit after imputation of missing data by the last observation carried forward method.
  The WBC counts were determined via complete blood count.
Time Frame: 30 months
Measure: Mean (Standard Deviation); unit: x10^6 cells/ml
Arm/Group | Control Group | GM-CSF Group
Number analyzed (Participants) | 9 | 9
x10^6 cells/ml
  Pre-WLL (Month -1) | 7.7 (1.8) | 6.2 (1.2)
  Baseline (Month 0) | 7.5 (1.7) | 8.7 (2.7)
  1 month | 6.8 (1.6) | 6.4 (1.6)
  3 months | 6.8 (1.4) | 5.9 (1.1)
  6 months | 6.8 (1.6) | 6.2 (1.3)
  10 months | 67 (1.8) | 6.1 (1.1)
  18 months | 6.8 (1.6) | 6.5 (10)
  30 months | 6.8 (1.6) | 6.1 (1.5)
Statistical Analysis 1: Comparison: Control Group vs GM-CSF Group; The secondary analysis includes evaluation of the difference in mean WBC counts between groups at the Pre-WLL visit after imputation of missing data using a last observation carried forward method; Test type: Superiority; p = 0.0582, t-test, 2 sided; Mean Difference (Final Values) = -1.55, 95% CI 2-sided [-3.17 to 0.06], Standard Error of Mean 0.78 — Calculated as the difference at the Pre-WLL visit in the mean WBC count in the GM-CSF Group minus the mean WBC count in the Control Group
Statistical Analysis 2: Comparison: Control Group vs GM-CSF Group; The secondary analysis includes evaluation of the difference in mean WBC counts between groups at the baseline visit after imputation of missing data using a last observation carried forward method; Test type: Superiority; p = 0.3068, t-test, 2 sided; Mean Difference (Final Values) = 1.15, 95% CI 2-sided [-1.17 to 3.48], Standard Error of Mean 1.09 — Calculated as the difference at the baseline visit in the mean WBC count in the GM-CSF Group minus the mean WBC count in the Control Group
Statistical Analysis 3: Comparison: Control Group vs GM-CSF Group; The secondary analysis includes evaluation of the difference in mean WBC counts between groups at the 1-month visit after imputation of missing data using a last observation carried forward method; Test type: Superiority; p = 0.5647, t-test, 2 sided; Mean Difference (Final Values) = -0.44, 95% CI 2-sided [-2.04 to 1.15], Standard Error of Mean 0.75 — Calculated as the difference at the 1-month visit in the mean WBC count in the GM-CSF Group minus the mean WBC count in the Control Group
Statistical Analysis 4: Comparison: Control Group vs GM-CSF Group; The secondary analysis includes evaluation of the difference in mean WBC counts between groups at the 3-month visit after imputation of missing data using a last observation carried forward method; Test type: Superiority; p = 0.1669, t-test, 2 sided; Mean Difference (Final Values) = -0.86, 95% CI 2-sided [-2.11 to 0.40], Standard Error of Mean 0.59 — Calculated as the difference at the 3-month visit in the mean WBC count in the GM-CSF Group minus the mean WBC count in the Control Group
Statistical Analysis 5: Comparison: Control Group vs GM-CSF Group; The secondary analysis includes evaluation of the difference in mean WBC counts between groups at the 6-month visit after imputation of missing data using a last observation carried forward method; Test type: Superiority; p = 0.4530, t-test, 2 sided; Mean Difference (Final Values) = -0.53, 95% CI 2-sided [-1.99 to 0.93], Standard Deviation 0.69 — Calculated as the difference at the 6-month visit in the mean WBC count in the GM-CSF Group minus the mean WBC count in the Control Group
Statistical Analysis 6: Comparison: Control Group vs GM-CSF Group; The secondary analysis includes evaluation of the difference in mean WBC counts between groups at the 10-month visit after imputation of missing data using a last observation carried forward method; Test type: Superiority; p = 0.4594, t-test, 2 sided; Mean Difference (Final Values) = -0.54, 95% CI 2-sided [-2.04 to 0.97], Standard Error of Mean 0.71 — Calculated as the difference at the 10-month visit in the mean WBC count in the GM-CSF Group minus the mean WBC count in the Control Group
Statistical Analysis 7: Comparison: Control Group vs GM-CSF Group; The secondary analysis includes evaluation of the difference in mean WBC counts between groups at the 18-month visit after imputation of missing data using a last observation carried forward method; Test type: Superiority; p = 0.6302, t-test, 2 sided; Mean Difference (Final Values) = -0.30, 95% CI 2-sided [-1.61 to 1.00], Standard Error of Mean 0.62 — Calculated as the difference at the 18-month visit in the mean WBC count in the GM-CSF Group minus the mean WBC count in the Control Group
Statistical Analysis 8: Comparison: Control Group vs GM-CSF Group; The secondary analysis includes evaluation of the difference in mean WBC counts between groups at the 30-month visit after imputation of missing data using a last observation carried forward method; Test type: Superiority; p = 0.3300, t-test, 2 sided; Mean Difference (Final Values) = -0.72, 95% CI 2-sided [-2.24 to 0.80], Standard Error of Mean 0.72 — Calculated as the difference at the 30-month visit in the mean WBC count in the GM-CSF Group minus the mean WBC count in the Control Group

13. Secondary Outcome: Between-Group Difference in Mean Platelet Counts
Description: Analysis Method: Between-group difference in platelet counts at each visit after imputation of missing data by the last observation carried forward method.
  The platelet counts were determined via complete blood count.
Time Frame: 30 months
Measure: Mean (Standard Deviation); unit: x10^6 cells/ml
Arm/Group | Control Group | GM-CSF Group
Number analyzed (Participants) | 9 | 9
x10^6 cells/ml
  Pre-WLL (Month -1) | 289 (96) | 236 (56)
  Baseline (Month 0) | 290 (111) | 269 (73)
  1 month | 266 (57) | 248 (46)
  3 months | 280 (83) | 252 (42)
  6 months | 267 (42) | 238 (45)
  10 months | 269 (50) | 242 (49)
  18 months | 263 (54) | 236 (42)
  30 months | 263 (53) | 232 (46)
Statistical Analysis 1: Comparison: Control Group vs GM-CSF Group; The secondary analysis includes evaluation of the difference in mean platelet counts between groups at the Pre-WLL visit after imputation of missing data using a last observation carried forward method; Test type: Superiority; p = 0.1864, t-test, 2 sided; Mean Difference (Final Values) = -53.72, 95% CI 2-sided [-136.4 to 28.96], Standard Error of Mean 38.79 — Calculated as the difference at the Pre-WLL visit in the mean platelet count in the GM-CSF Group minus the mean platelet count in the Control Group
Statistical Analysis 2: Comparison: Control Group vs GM-CSF Group; The secondary analysis includes evaluation of the difference in mean platelet counts between groups at the baseline visit after imputation of missing data using a last observation carried forward method; Test type: Superiority; p = 0.6541, t-test, 2 sided; Mean Difference (Final Values) = -21.17, 95% CI 2-sided [-119.8 to 77.51], Standard Error of Mean 46.30 — Calculated as the difference at the baseline visit in the mean platelet count in the GM-CSF Group minus the mean platelet count in the Control Group
Statistical Analysis 3: Comparison: Control Group vs GM-CSF Group; The secondary analysis includes evaluation of the difference in mean platelet counts between groups at the 1-month visit after imputation of missing data using a last observation carried forward method; Test type: Superiority; p = 0.4560, t-test, 2 sided; Mean Difference (Final Values) = -18.78, 95% CI 2-sided [-70.89 to 33.33], Standard Error of Mean 24.58 — Calculated as the difference at the 1-month visit in the mean platelet count in the GM-CSF Group minus the mean platelet count in the Control Group
Statistical Analysis 4: Comparison: Control Group vs GM-CSF Group; The secondary analysis includes evaluation of the difference in mean platelet counts between groups at the 3-month visit after imputation of missing data using a last observation carried forward method; Test type: Superiority; p = 0.3721, t-test, 2 sided; Mean Difference (Final Values) = -28.44, 95% CI 2-sided [-94.12 to 37.23], Standard Error of Mean 30.98 — Calculated as the difference at the 3-month visit in the mean platelet count in the GM-CSF Group minus the mean platelet count in the Control Group
Statistical Analysis 5: Comparison: Control Group vs GM-CSF Group; The secondary analysis includes evaluation of the difference in mean platelet counts between groups at the 6-month visit after imputation of missing data using a last observation carried forward method; Test type: Superiority; p = 0.1812, t-test, 2 sided; Mean Difference (Final Values) = -28.78, 95% CI 2-sided [-72.41 to 14.86], Standard Error of Mean 20.58 — Calculated as the difference at the 6-month visit in the mean platelet count in the GM-CSF Group minus the mean platelet count in the Control Group
Statistical Analysis 6: Comparison: Control Group vs GM-CSF Group; The secondary analysis includes evaluation of the difference in mean platelet counts between groups at the 10-month visit after imputation of missing data using a last observation carried forward method; Test type: Superiority; p = 0.2805, t-test, 2 sided; Mean Difference (Final Values) = -26.11, 95% CI 2-sided [-75.67 to 23.44], Standard Error of Mean 23.38 — Calculated as the difference at the 10-month visit in the mean platelet count in the GM-CSF Group minus the mean platelet count in the Control Group
Statistical Analysis 7: Comparison: Control Group vs GM-CSF Group; The secondary analysis includes evaluation of the difference in mean platelet counts between groups at the 18-month visit after imputation of missing data using a last observation carried forward method; Test type: Superiority; p = 0.2470, t-test, 2 sided; Mean Difference (Final Values) = -27.33, 95% CI 2-sided [-75.56 to 20.89], Standard Error of Mean 22.75 — Calculated as the difference at the 18-month visit in the mean platelet count in the GM-CSF Group minus the mean platelet count in the Control Group
Statistical Analysis 8: Comparison: Control Group vs GM-CSF Group; The secondary analysis includes evaluation of the difference in mean platelet counts between groups at the 30-month visit after imputation of missing data using a last observation carried forward method; Test type: Superiority; p = 0.2070, t-test, 2 sided; Mean Difference (Final Values) = -31.00, 95% CI 2-sided [-80.97 to 18.97], Standard Error of Mean 23.57 — Calculated as the difference at the 30-month visit in the mean platelet count in the GM-CSF Group minus the mean platelet count in the Control Group

14. Secondary Outcome: Between-Group Difference in Mean 36-Item Short Form Survey (SF-36) General Health Score
Description: Primary Analysis: Between-group difference in mean SF-36 General Health Score at each study visit after the scheduled baseline WLL was evaluated using repeated measures analysis of variance (ANOVA) after adjustment for baseline values, gender, age, and the number of patients at risk at each time point.
  Secondary analysis: Between-group difference in SF-36 General Health Score at each visit after imputation of missing data by the last observation carried forward method.
  The SF-36 General Health Score were determined from the RAND 36-Item Health Survey. Scoring the SF-36 questionnaire is a two-step process. First, pre-coded numeric values are recoded per the scoring key. All items are scored on a scale of 0 to 100 so that a high score defines a more favorable health state. Scores represent the percentage of total possible score achieved. In step 2, General Health is determined from the average score for questions 1, 33, 34, 35, and 36.
Time Frame: 30 months
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Control Group | GM-CSF Group
Number analyzed (Participants) | 9 | 9
Score on a scale
  Pre-WLL (Month -1) | 44 (27) | 39 (22)
  1 month | 77 (20) | 85 (15)
  3 months | 79 (18) | 93 (6.1)
  6 months | 77 (22) | 95 (4.3)
  10 months | 72 (26) | 84 (15)
  18 months | 74 (26) | 84 (18)
  30 months | 71 (28) | 88 (8.7)
Statistical Analysis 1: Comparison: Control Group vs GM-CSF Group; Primary analysis; Test type: Superiority; p = 0.1490, Repeated measures ANOVA; [statistical method as in outcome 3, analysis 1]; Mean Difference (Final Values) = 4.72, 95% CI 2-sided [-1.88 to 11.33] — Calculated as the difference in the mean value of the SF-36 General Health Score in the GM-CSF Group minus the Control Group
Statistical Analysis 2: Comparison: Control Group vs GM-CSF Group; The secondary analysis includes evaluation of the difference in mean SF-36 General Health Score between groups at the Pre-WLL visit after imputation of missing data using a last observation carried forward method; Test type: Superiority; p = 0.7263, t-test, 2 sided; Mean Difference (Final Values) = -4.31, 95% CI 2-sided [-30.04 to 21.43], Standard Error of Mean 12.07 — Calculated as the difference at the Pre-WLL visit in the mean SF-36 General Health Score in the GM-CSF Group minus the mean SF-36 General Health Score in the Control Group
Statistical Analysis 3: Comparison: Control Group vs GM-CSF Group; The secondary analysis includes evaluation of the difference in SF-36 General Health Score between groups at the 1-month visit after imputation of missing data using a last observation carried forward method; Test type: Superiority; p = 0.3298, t-test, 2 sided; Mean Difference (Final Values) = 8.33, 95% CI 2-sided [-9.24 to 25.91], Standard Error of Mean 8.29 — Calculated as the difference at the 1-month visit in the mean SF-36 General Health Score in the GM-CSF Group minus the mean SF-36 General Health Score in the Control Group
Statistical Analysis 4: Comparison: Control Group vs GM-CSF Group; The secondary analysis includes evaluation of the difference in SF-36 General Health Score between groups at the 3-month visit after imputation of missing data using a last observation carried forward method; Test type: Superiority; p = 0.0478, t-test, 2 sided; Mean Difference (Final Values) = 13.89, 95% CI 2-sided [-0.15 to 27.62], Standard Error of Mean 6.48 — Calculated as the difference at the 3-month visit in the mean SF-36 General Health Score in the GM-CSF Group minus the mean SF-36 General Health Score in the Control Group
Statistical Analysis 5: Comparison: Control Group vs GM-CSF Group; The secondary analysis includes evaluation of the difference in mean SF-36 General Health Score between groups at the 6-month visit after imputation of missing data using a last observation carried forward method; Test type: Superiority; p = 0.0281, t-test, 2 sided; Mean Difference (Final Values) = 17.78, 95% CI 2-sided [2.16 to 33.39], Standard Error of Mean 7.37 — Calculated as the difference at the 6-month visit in the mean SF-36 General Health Score in the GM-CSF Group minus the mean SF-36 General Health Score in the Control Group
Statistical Analysis 6: Comparison: Control Group vs GM-CSF Group; The secondary analysis includes evaluation of the difference in mean SF-36 General Health Score between groups at the 10-month visit after imputation of missing data using a last observation carried forward method; Test type: Superiority; p = 0.2634, t-test, 2 sided; Mean Difference (Final Values) = 11.67, 95% CI 2-sided [-9.67 to 33.00], Standard Error of Mean 10.07 — Calculated as the difference at the 10-month visit in the mean SF-36 General Health Score in the GM-CSF Group minus the mean SF-36 General Health Score in the Control Group
Statistical Analysis 7: Comparison: Control Group vs GM-CSF Group; The secondary analysis includes evaluation of the difference in mean SF-36 General Health Score between groups at the 18-month visit after imputation of missing data using a last observation carried forward method; Test type: Superiority; p = 0.3548, t-test, 2 sided; Mean Difference (Final Values) = 10.00, 95% CI 2-sided [-12.24 to 32.24], Standard Error of Mean 10.49 — Calculated as the difference at the 18-month visit in the mean SF-36 General Health Score in the GM-CSF Group minus the mean SF-36 General Health Score in the Control Group
Statistical Analysis 8: Comparison: Control Group vs GM-CSF Group; The secondary analysis includes evaluation of the difference in mean SF-36 General Health Score between groups at the 30-month visit after imputation of missing data using a last observation carried forward method; Test type: Superiority; p = 0.1043, t-test, 2 sided; Mean Difference (Final Values) = 16.67, 95% CI 2-sided [-3.85 to 37.18], Standard Error of Mean 9.68 — Calculated as the difference at the 30-month visit in the mean SF-36 General Health Score in the GM-CSF Group minus the mean SF-36 General Health Score in the Control Group

ADVERSE EVENTS:
Time Frame: Adverse events, serious adverse events, adverse drug reactions, and adverse events leading to treatment discontinuation, including clinically significant changes in laboratory tests, during the 30 months immediately following administration of the scheduled baseline bilateral WLL at Study Month 0 were collected.
Arm/Group | Control Group | GM-CSF Group
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 0/9 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No